CLINICAL TRIAL: NCT02472496
Title: Korean Coronary Overlapping Stenting Registy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Dong-Bin Kim, Professor, The Catholic University of Korea
Other Study IDs: 5-2013-B0001-00245
Record Dates: First submitted 2015-06-10; First posted 2015-06-16 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Korean Coronary Overlapping Stenting Registry is a multicenter database which includes percutaneous intervention using drug-eluting stents from cardiovascular centers in eight affiliated hospitals of The Catholic University of Korea

DETAILED DESCRIPTION:
The Korean Coronary Overlapping Stenting Registry is a multi-center, real-world of drug-eluting stent overlap.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Drug-eluting stent overlap

Exclusion Criteria:

* Overlap with previous stent
* Cardiogenic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary lesion treated with overlapping drug-eluting stents
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of the composite outcomes of cardiac death, myocardial infarction, and target lesion revascularization | 3 years

SECONDARY OUTCOMES:
Cardiac death | 3 years
Myocardial infarction | 3 years
Target lesion revascularization | 3 years
stent thrombosis | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Bin Kim, MD, Principal Investigator — The Catholic University of Korea
Locations (1):
- Korea cardiovascular center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raber L, Juni P, Loffel L, Wandel S, Cook S, Wenaweser P, Togni M, Vogel R, Seiler C, Eberli F, Luscher T, Meier B, Windecker S. Impact of stent overlap on angiographic and long-term clinical outcome in patients undergoing drug-eluting stent implantation. J Am Coll Cardiol. 2010 Mar 23;55(12):1178-1188. doi: 10.1016/j.jacc.2009.11.052. PMID 20298923